CLINICAL TRIAL: NCT02782858
Title: An International, Double-blind, Randomised, Placebo-controlled Phase IIb Trial to Assess the Efficacy, Safety, and Pharmacokinetics of GNbAC1 in Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: Clinical Trial Assessing the HERV-W Env Antagonist GNbAC1 for Efficacy in MS
Acronym: CHANGE-MS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GeNeuro SA (Industry)
Collaborators: Les Laboratoires Servier (LLS) (Unknown); Institut de Recherches Internationales Servier (Other); Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNC-003; 2015-004059-29 (EudraCT Number)
Record Dates: First submitted 2016-05-23; First posted 2016-05-25 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2018-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Multiple Sclerosis Relapsing-Remitting; GNbAC1; MRI; Monoclonal antibody; Multiple Sclerosis associated retrovirus MSRV; MS; RRMS; HERV-W; Temelimab
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — temelimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose 1 GNbAC1 (Experimental): Monthly IV repeated dose
  Interventions: Drug: GNbAC1
- Dose 2 GNbAC1 (Experimental): Monthly IV repeated dose
  Interventions: Drug: GNbAC1
- Dose 3 GNbAC1 (Experimental): Monthly IV repeated dose
  Interventions: Drug: GNbAC1
- Placebo (Placebo Comparator): Monthly IV repeated dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GNbAC1 — Monthly IV repeated dose
  Arms: Dose 1 GNbAC1; Dose 2 GNbAC1; Dose 3 GNbAC1
Drug: Placebo — Monthly IV repeated dose
  Arms: Placebo

SUMMARY:
The humanised IgG4 monoclonal antibody GNbAC1 targets the envelope protein (Env) of the human endogenous multiple sclerosis-associated retrovirus (HERV-W MSRV), which may play a critical role in multiple sclerosis (MS).

This study evaluates the effect on MRI lesions parameters, the safety and pharmacokinetics of GNbAC1 in patients with relapsing remitting multiple sclerosis.

ELIGIBILITY:
Main Inclusion Criteria:

* For male or female with reproductive potential, use of reliable means of contraception;
* RRMS according to the 2010 revised McDonald criteria;
* Disease activity characterised by at least one documented relapse within the last 12 months and /or at least one Gd-enhancing T1 lesion at selection or evidenced within the last 3 months;
* EDSS score < 6.0.

Main Exclusion Criteria:

* Patients suffering from Secondary Progressive MS and Primary Progressive MS at screening;
* Pregnant and nursing women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cumulative number of Gd-enhancing T1 lesions in brain MRI | Week 12 to 24

CONTACTS AND LOCATIONS:
Locations (12):
- Sofia, Bulgaria
- Zagreb, Croatia
- Jihlava, Czechia
- Tallinn, Estonia
- Berlin, Germany
- Budapest, Hungary
- Roma, Italy
- Warsaw, Poland
- Moscow, Russia
- Belgrade, Serbia
- Barcelona, Spain
- Kharkiv, Ukraine

REFERENCES:
- [Derived] Hartung HP, Derfuss T, Cree BA, Sormani MP, Selmaj K, Stutters J, Prados F, MacManus D, Schneble HM, Lambert E, Porchet H, Glanzman R, Warne D, Curtin F, Kornmann G, Buffet B, Kremer D, Kury P, Leppert D, Ruckle T, Barkhof F. Efficacy and safety of temelimab in multiple sclerosis: Results of a randomized phase 2b and extension study. Mult Scler. 2022 Mar;28(3):429-440. doi: 10.1177/13524585211024997. Epub 2021 Jul 9. PMID 34240656